CLINICAL TRIAL: NCT03439280
Title: A Phase 1/2a Open-label, Dose-Escalation Study to Investigate the Safety and Tolerability, Efficacy, Pharmacokinetics, and Immunogenicity of TAK-079 Administered Subcutaneously as a Single Agent in Patients With Relapsed/Refractory Multiple Myeloma
Brief Title: A Study to Investigate the Safety, Tolerability, Efficacy, Pharmacokinetics, and Immunogenicity of TAK-079 Administered Subcutaneously as a Single Agent in Participants With Relapsed/Refractory (r/r) Multiple Myeloma (MM)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TAK-079-1501; U1111-1208-3202 (Other: WHO)
Record Dates: First submitted 2018-02-14; First posted 2018-02-20 (Actual); Results first posted 2023-02-24 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-01

CONDITIONS: Relapsed/Refractory; Multiple Myeloma
Keywords: Drug therapy, TAK-079, pomalidomide and dexamethasone, CD38 monoclonal antibody
MeSH Terms: conditions — Recurrence; Multiple Myeloma | interventions — pomalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Phase 1 Dose Escalation Cohort: Mezagitamab 45 mg (Experimental): Mezagitamab 45 mg, subcutaneously (SC), once weekly for 8 weeks, then once every 2 weeks for 16 weeks, and then once every 4 weeks thereafter in a 28-day treatment cycle until progressive disease (PD), unacceptable toxicities or withdrawal due to other reasons.
  Interventions: Drug: Mezagitamab
- Phase 1 Dose Escalation Cohort: Mezagitamab 135 mg (Experimental): Mezagitamab 135 mg, SC, once weekly for 8 weeks, then once every 2 weeks for 16 weeks, and then once every 4 weeks thereafter in a 28-day treatment cycle until PD, unacceptable toxicities or withdrawal due to other reasons.
  Interventions: Drug: Mezagitamab
- Phase 1 Dose Escalation Cohort: Mezagitamab 300 mg (Experimental): Mezagitamab 300 mg, SC, once weekly for 8 weeks, then once every 2 weeks for 16 weeks, and then once every 4 weeks thereafter in a 28-day treatment cycle until PD, unacceptable toxicities or withdrawal due to other reasons.
  Interventions: Drug: Mezagitamab
- Phase 1 Dose Escalation Cohort: Mezagitamab 600 mg (Experimental): Mezagitamab 600 mg, SC, once weekly for 8 weeks, then once every 2 weeks for 16 weeks, and then once every 4 weeks thereafter in a 28-day treatment cycle until PD, unacceptable toxicities or withdrawal due to other reasons.
  Interventions: Drug: Mezagitamab
- Phase 1 Dose Escalation Cohort: Mezagitamab 1200 mg (Experimental): Mezagitamab 1200 mg, SC, once weekly for 8 weeks, then once every 2 weeks for 16 weeks, and then once every 4 weeks thereafter in a 28-day treatment cycle until PD, unacceptable toxicities or withdrawal due to other reasons.
  Interventions: Drug: Mezagitamab
- Phase 1 Combination Cohort: Mezagitamab 300 mg + PomDex (Experimental): Mezagitamab 300 mg, SC, once weekly for 8 weeks, then once every 2 weeks for 16 weeks, and then once every 4 weeks thereafter along with pomalidomide, at product-labelled dose, orally, once daily on Days 1 to 21 and dexamethasone, at product-labelled dose, orally, once on Days 1, 8, 15, and 22 in a 28-day treatment cycle until PD.
  Interventions: Drug: Mezagitamab; Drug: Pomalidomide; Drug: Dexamethasone
- Phase 2a: Mezagitamab (Experimental): Mezagitamab, SC, once weekly for 8 weeks, then once every 2 weeks for 16 weeks, and then once every 4 weeks thereafter in a 28-day treatment cycle until PD, unacceptable toxicities or withdrawal due to other reasons. TAK-079 dose for this phase was to be determined based on review of the available safety, efficacy, pharmacokinetic, and pharmacodynamic data obtained from the Phase 1 portion of the study. However, Phase 2a of the study was not opened for enrollment due to changes in the Sponsor's overall clinical development plan.
  Interventions: Drug: Mezagitamab

INTERVENTIONS:
Drug: Mezagitamab — Mezagitamab subcutaneously.
  Other Names: TAK-079
Drug: Pomalidomide — Pomalidomide orally.
  Arms: Phase 1 Combination Cohort: Mezagitamab 300 mg + PomDex
Drug: Dexamethasone — Dexamethasone orally.
  Arms: Phase 1 Combination Cohort: Mezagitamab 300 mg + PomDex

SUMMARY:
The purpose of this study is to assess the safety and tolerability, maximum tolerated dose (MTD)/recommended phase 2 dose (RP2D) of TAK-079 monotherapy and when combined with a backbone regimen of pomalidomide and dexamethasone (PomDex) in Phase 1, and to provide a preliminary evaluation of the clinical activity of TAK-079 monotherapy in Phase 2a in participants with r/r MM.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-079. TAK-079 is being tested to treat people who have relapsed and/or refractory multiple myeloma (RRMM). This study will assess the safety, tolerability, efficacy, pharmacokinetics, and immunogenicity of TAK-079 monotherapy and will provide a preliminary assessment of its activity against MM. The study is designed to consist of 2 phases: Phase 1 and Phase 2a.

The study could enroll approximately 100 participants. The study population of Phase 1 will consist of approximately 55 participants. Participants in Phase 1 will be assigned to TAK-079 and dose-escalation will range from 45 mg to 1800 mg.

The study population of Phase 2a will consist of approximately 48 participants. Dose for Phase 2a will be based upon review of the available safety, efficacy, pharmacokinetic, and pharmacodynamic data from the preceding cohorts of Phase 1.

This multi-center trial will be conducted in the United States. The overall time to participate in this study is 42 months (3.5 years). In Phase 1, participants who stop treatment for any other reason other than PD will continue to have progression-free survival (PFS) follow-up at the site every 4 weeks from the last dose of study drug up to 12 months or until PD, death, loss to follow-up, consent withdrawal or study termination. Participants will be followed 30 days after last dose of study drug or until the start of subsequent alternative anti-cancer therapy, whichever occurs first, for a follow up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Eastern Cooperative Oncology Group (ECOG) performance status of <=2.
2. Has received previous myeloma-specific therapy.
3. In the Combination Cohort (TAK-079-PomDex) only must be able to take concurrent prophylactic anticoagulation per standard clinical practice as directed by the investigator and the Pomalyst product information.
4. Documentation of RRMM as defined by the International Myeloma Working Group (IMWG) criteria.
5. For Participants with MM, measurable disease defined as one of the following:

   * Serum M-protein >=0.5 g/dL (>=5 gram per liter [g/L]).
   * Urine M-protein >=200 mg/24 hours.
   * In participants without measurable M-protein in serum protein electrophoresis (SPEP) or urine protein electrophoresis (UPEP), a serum FLC assay result with involved FLC level >=10 mg/dL (>=100 milligram per liter [mg/L]), provided serum FLC ratio is abnormal.
6. Prior therapy should meet all the following criteria:

   Participants in the dose Escalation Cohort (escalation phase) and participants in the dose Confirmation Cohort;
   * Should be previously treated with at least a proteasome inhibitor (PI), an immunomodulatory drug (IMiD), and a steroid. Note: Participants who have had a previous autologous stem cell transplant will have additionally been exposed to an alkylating agent; however, participant who have not had a previous autologous stem cell transplant may not have been exposed to an alkylating agent per standard practice.
   * Should be refractory or intolerant to at least 1 PI and at least 1 IMiD.
   * Should either have received >= 3 prior lines of therapy or should have received at least 2 prior lines of therapy if one of those lines included a combination of PI and IMiD.
   * In phase 1, previous exposure to an anti-CD38 agent, as a single agent or in combination, is allowed but is not required. (Participants in the dose Escalation Cohort).
   * In phase 1 dose Confirmation Cohort, cohorts of participants that are refractory at any time to at least 1 anti-CD38 agent or who are anti-CD38 naïve will be enrolled.

   Participants in the Combination Cohort (TAK-079 added to PomDex cohort only):
   * Have undergone prior therapy with >=2 prior anti-myeloma therapies (line of therapy defined below).
   * Has either relapsed or relapsed and refractory disease. Should have progressed on or within 60 days of completing the last anti-myeloma therapy (refractory defined below).
7. In the phase 2a portion of the study, up to 2 cohorts of participants with RRMM may be enrolled: 1 that is refractory to at least 1 anti-CD38 monoclonal antibody (mAb) therapy at any time during treatment and 1 that is naïve to daratumumab.

Note:

o Refractory is defined as at least a 25% increase in M-protein (response of stable disease during prior therapy) or PD during treatment or within 60 days after last dose of prior therapy.

Exclusion Criteria:

1. Sensory or motor neuropathy of National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Grade >=3.
2. Have received allogeneic stem cell transplant.
3. Have received anti-CD38 antibody therapy and do not fulfill a 180-day washout period before receiving TAK-079.
4. Not recovered from adverse reactions to prior myeloma treatment or procedures (chemotherapy, immunotherapy, radiation therapy) to NCI CTCAE Grade <=1 or baseline, excluding alopecia.
5. Clinical signs of central nervous system (CNS) involvement of MM.
6. Active chronic hepatitis B virus (HBV) or hepatitis C virus (HCV) infection, active HIV, or cytomegalovirus (CMV) infection.
7. POEMS (polyneuropathy, organomegaly, endocrinopathy, monoclonal gammopathy and skin changes) syndrome, monoclonal gammopathy of unknown significance, smoldering myeloma, solitary plasmacytoma, amyloidosis, Waldenström macroglobulinemia, or IgM myeloma.
8. Positive Coombs tests at screening.
9. For participants in the Combination Cohort (TAK-079-PomDex) only: participant has previously received pomalidomide or has hypersensitivity to thalidomide or lenalidomide.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-04-20 (Actual); Primary Completion 2022-01-28 (Actual); Study Completion 2022-01-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (7):
- United States (7):
  - City of Hope - Duarte, Duarte, California
  - Washington University School of Medicine, St Louis, Missouri
  - Mount Sinai Hospital-The Donald H. Ruttenberg Cancer Treatment Center, New York, New York
  - Weill Cornell Medical Center, Div. of Hematology Medical Oncology, New York, New York
  - Oregon Health & Science University Knight Cancer Institute, Portland, Oregon
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Krishnan AY, Patel KK, Mohan M, Jagannath S, Niesvizky R, Silbermann RW, Yu Z, Long T, McDonnell SRP, Berg D, Stockerl-Goldstein KE. Phase 1b study of the anti-CD38 antibody mezagitamab in patients with relapsed/refractory multiple myeloma. Blood Neoplasia. 2024 Sep 18;1(4):100043. doi: 10.1016/j.bneo.2024.100043. eCollection 2024 Dec. PMID 40552138

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 7 investigative sites in the United States from 20 April 2018 to 28 January 2022.
Pre-assignment Details: Participants with a diagnosis of relapsed or refractory (R/R) multiple myeloma (MM) were enrolled in Phase 1 to receive mezagitamab in a dose escalating manner and in combination with PomDex. Phase 2a of the study was not opened for enrollment due to changes in the Sponsor's overall clinical development plan.
Period: Overall Study
Arm/Group | Phase 1 Dose Escalation Cohort: Mezagitamab 45 mg | Phase 1 Dose Escalation Cohort: Mezagitamab 135 mg | Phase 1 Dose Escalation Cohort: Mezagitamab 300 mg | Phase 1 Dose Escalation Cohort: Mezagitamab 600 mg | Phase 1 Dose Escalation Cohort: Mezagitamab 1200 mg | Phase 1 Combination Cohort: Mezagitamab 300 mg + PomDex | Phase 2a: Mezagitamab
Started | 4 | 3 | 12 | 22 | 3 | 6 | 0
Completed | 4 | 3 | 12 | 22 | 3 | 6 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All-enrolled analysis set included all participants enrolled into the study, regardless of whether they received any dose of study drug.
Groups:
- Phase 1 Dose Escalation Cohort: Mezagitamab 45 mg: Mezagitamab 45 mg, SC, once weekly for 8 weeks, then once every 2 weeks for 16 weeks, and then once every 4 weeks thereafter in a 28-day treatment cycle until PD, unacceptable toxicities or withdrawal due to other reasons.
- Total: Total of all reporting groups
Arm/Group | Phase 1 Dose Escalation Cohort: Mezagitamab 45 mg | Phase 1 Dose Escalation Cohort: Mezagitamab 135 mg | Phase 1 Dose Escalation Cohort: Mezagitamab 300 mg | Phase 1 Dose Escalation Cohort: Mezagitamab 600 mg | Phase 1 Dose Escalation Cohort: Mezagitamab 1200 mg | Phase 1 Combination Cohort: Mezagitamab 300 mg + PomDex | Total
Number analyzed (Participants) | 4 | 3 | 12 | 22 | 3 | 6 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.3 (9.71) | 69.0 (5.00) | 67.3 (5.99) | 69.3 (7.59) | 62.0 (11.14) | 64.2 (8.50) | 67.3 (7.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 2 | 8 | 0 | 4 | 17
  Male | 2 | 2 | 10 | 14 | 3 | 2 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2 | 3 | 1 | 0 | 8
  Not Hispanic or Latino | 2 | 3 | 10 | 19 | 2 | 5 | 41
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 0 | 3 | 0 | 2 | 9
  White | 1 | 0 | 9 | 15 | 3 | 3 | 31
  More than one race | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 1 | 1 | 1 | 3 | 0 | 1 | 7
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 3 | 12 | 22 | 3 | 6 | 50

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Number of Participants Reporting One or More Treatment-emergent Adverse Events (TEAEs)
Description: TEAEs were any untoward medical occurrence (called an adverse event [AE]) that occurred after administration of the first dose of any study drug and through 30 days after the last dose of any study drug.
Time Frame: From the first dose of study drug through 30 days after the last dose (up to approximately 3.7 years)
Population: Safety analysis set included all enrolled participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 Dose Escalation Cohort: Mezagitamab 45 mg | Phase 1 Dose Escalation Cohort: Mezagitamab 135 mg | Phase 1 Dose Escalation Cohort: Mezagitamab 300 mg | Phase 1 Dose Escalation Cohort: Mezagitamab 600 mg | Phase 1 Dose Escalation Cohort: Mezagitamab 1200 mg | Phase 1 Combination Cohort: Mezagitamab 300 mg + PomDex
Number analyzed (Participants) | 4 | 3 | 12 | 22 | 3 | 6
Participants | 4 | 3 | 12 | 22 | 3 | 6

2. Primary Outcome: Phase 1: Number of Participants With Dose-limiting Toxicities (DLTs)
Description: DLTs were defined as any of the following events: Grade 4 laboratory abnormalities, except those events that were clearly due to extraneous causes; nonhematologic TEAEs of grade greater than or equal to (>=3) except grade 3 nausea/vomiting, fatigue lasting less than 72 hours, elevation of alanine aminotransferase (ALT) or aspartate aminotransferase (AST) that resolves to grade less than or equal to (<=)1 or baseline within 7 days, injection reaction (IR) that responds to symptomatic treatment; Hematologic TEAEs of National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) grade >=4, except grade >=3 hemolysis, grade 3 low platelet or higher count with clinically meaningful bleeding; and an incomplete recovery from treatment-related toxicity causing a greater than (>) 2-week delay in the next scheduled injection before the initiation of Cycle 2 will be considered a DLT.
Time Frame: Cycle 1 (cycle length=28 days)
Population: DLT-evaluable analysis set included participants who received all Cycle 1 doses of mezagitamab and completed Cycle 1 procedures or experienced a DLT in Cycle 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 Dose Escalation Cohort: Mezagitamab 45 mg | Phase 1 Dose Escalation Cohort: Mezagitamab 135 mg | Phase 1 Dose Escalation Cohort: Mezagitamab 300 mg | Phase 1 Dose Escalation Cohort: Mezagitamab 600 mg | Phase 1 Dose Escalation Cohort: Mezagitamab 1200 mg | Phase 1 Combination Cohort: Mezagitamab 300 mg + PomDex
Number analyzed (Participants) | 4 | 3 | 10 | 17 | 3 | 4
Participants | 0 | 0 | 0 | 0 | 0 | 1

3. Primary Outcome: Phase 1: Number of Participants With Grade 3 or Higher TEAEs
Description: AE Grades were evaluated as per National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 4.03. Grade 3 scaled as severe or medically significant but not immediately life-threatening; Grade 4 scaled as life-threatening consequences; and Grade 5 scaled as death related to AE.
Time Frame: From the first dose of study drug through 30 days after the last dose (up to approximately 3.7 years)
Population: Safety analysis set included all enrolled participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 Dose Escalation Cohort: Mezagitamab 45 mg | Phase 1 Dose Escalation Cohort: Mezagitamab 135 mg | Phase 1 Dose Escalation Cohort: Mezagitamab 300 mg | Phase 1 Dose Escalation Cohort: Mezagitamab 600 mg | Phase 1 Dose Escalation Cohort: Mezagitamab 1200 mg | Phase 1 Combination Cohort: Mezagitamab 300 mg + PomDex
Number analyzed (Participants) | 4 | 3 | 12 | 22 | 3 | 6
Participants | 2 | 1 | 3 | 12 | 1 | 6

4. Primary Outcome: Phase 1: Number of Participants With Serious TEAEs
Description: TEAEs were any untoward medical occurrence (called an AE) that occurred after administration of the first dose of any study drug and through 30 days after the last dose of any study drug. A SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; or congenital anomaly; or a medically important event.
Time Frame: From the first dose of study drug through 30 days after the last dose (up to approximately 3.7 years)
Population: Safety analysis set included all enrolled participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 Dose Escalation Cohort: Mezagitamab 45 mg | Phase 1 Dose Escalation Cohort: Mezagitamab 135 mg | Phase 1 Dose Escalation Cohort: Mezagitamab 300 mg | Phase 1 Dose Escalation Cohort: Mezagitamab 600 mg | Phase 1 Dose Escalation Cohort: Mezagitamab 1200 mg | Phase 1 Combination Cohort: Mezagitamab 300 mg + PomDex
Number analyzed (Participants) | 4 | 3 | 12 | 22 | 3 | 6
Participants | 0 | 0 | 1 | 8 | 1 | 2

5. Primary Outcome: Phase 1: Number of Participants With TEAEs Leading to Treatment Discontinuation
Description: TEAEs leading to discontinuation were any untoward medical occurrence (called an AE) that occurred after administration of the first dose of any study drug and through 30 days after the last dose of any study drug leading to discontinuation of any of the study treatment when given in combination.
Time Frame: From the first dose of study drug through 30 days after the last dose (up to approximately 3.7 years)
Population: Safety analysis set included all enrolled participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 Dose Escalation Cohort: Mezagitamab 45 mg | Phase 1 Dose Escalation Cohort: Mezagitamab 135 mg | Phase 1 Dose Escalation Cohort: Mezagitamab 300 mg | Phase 1 Dose Escalation Cohort: Mezagitamab 600 mg | Phase 1 Dose Escalation Cohort: Mezagitamab 1200 mg | Phase 1 Combination Cohort: Mezagitamab 300 mg + PomDex
Number analyzed (Participants) | 4 | 3 | 12 | 22 | 3 | 6
Participants | 0 | 0 | 0 | 2 | 0 | 3

6. Primary Outcome: Phase 1: Number of Participants With TEAEs Leading to Dose Modifications
Description: TEAEs were any untoward medical occurrence (called an AE) that occurred after administration of the first dose of any study drug and through 30 days after the last dose of any study drug. Dose modification includes dose delayed, reduced, and drug discontinued permanently. Dose reduced includes scenarios where the dose was skipped, held, or missed. Dose modifications also refer to a modification of any drug in the study treatment when given in combination.
Time Frame: From the first dose of study drug through 30 days after the last dose (up to approximately 3.7 years)
Population: Safety analysis set included all enrolled participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 Dose Escalation Cohort: Mezagitamab 45 mg | Phase 1 Dose Escalation Cohort: Mezagitamab 135 mg | Phase 1 Dose Escalation Cohort: Mezagitamab 300 mg | Phase 1 Dose Escalation Cohort: Mezagitamab 600 mg | Phase 1 Dose Escalation Cohort: Mezagitamab 1200 mg | Phase 1 Combination Cohort: Mezagitamab 300 mg + PomDex
Number analyzed (Participants) | 4 | 3 | 12 | 22 | 3 | 6
Participants | 1 | 1 | 1 | 11 | 1 | 6

7. Primary Outcome: Phase 2a: Overall Response Rate (ORR)
Description: ORR is defined as the percentage of participants who achieved a partial response (PR) better during the study. PR is defined as >=50% reduction of serum M-protein and reduction in 24-hour urinary M-protein by >= 90% or to < 200 milligram per (mg/) 24 hours. If serum and urine M protein are not measurable, >= 50% decrease in difference between involved and uninvolved free light chain (FLC) levels is required in place of M protein criteria.
Time Frame: Up to approximately 3.7 years
Population: Data was not collected as Phase 2a of the study was not opened for enrollment due to changes in the Sponsor's overall clinical development plan.
Arm/Group | Phase 2a: Mezagitamab
Number analyzed (Participants) | 0

8. Secondary Outcome: Cmax: Maximum Observed Serum Concentration for TAK-079
Time Frame: Cycles 1 and 2: Day 1 pre-dose and at multiple time points (up to 168 hours) post-dose (cycle length=28 days)
Population: Pharmacokinetic (PK) analysis set included those participants from the safety analysis set who had sufficient dosing data and mezagitamab concentration-time data to permit the calculation of PK parameters. Number analyzed is the number of participants with data available for analysis at the given timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Phase 1 Dose Escalation Cohort: Mezagitamab 45 mg | Phase 1 Dose Escalation Cohort: Mezagitamab 135 mg | Phase 1 Dose Escalation Cohort: Mezagitamab 300 mg | Phase 1 Dose Escalation Cohort: Mezagitamab 600 mg | Phase 1 Dose Escalation Cohort: Mezagitamab 1200 mg | Phase 1 Combination Cohort: Mezagitamab 300 mg + PomDex
Number analyzed (Participants) | 4 | 3 | 12 | 22 | 3 | 6
nanograms per milliliter (ng/mL)
  Cycle 1 Week 1 | 47.0 (1908.7) | 1660 (460.1) | 5810 (599.9) | 21300 (196.6) | 46000 (58.0) | 5690 (223.5)
  Cycle 2 Week 1: number analyzed (Participants) | 4 | 3 | 11 | 16 | 3 | 6
  Cycle 2 Week 1 | 228 (4373.4) | 12900 (142.3) | 42700 (86.3) | 143000 (66.2) | 174000 (76.3) | 25800 (69.8)

9. Secondary Outcome: Tmax: Time to Reach the Maximum Observed Serum Concentration (Cmax) for TAK-079
Time Frame: Cycles 1 and 2: Day 1 pre-dose and at multiple time points (up to 190.95 hours) post-dose (cycle length=28 days)
Population: PK analysis set included those participants from the safety analysis set who had sufficient dosing data and mezagitamab concentration-time data to permit the calculation of PK parameters. Number analyzed is the number of participants with data available for analysis at the given timepoint.
Measure: Median (Full Range); unit: hours (h)
Groups:
- Phase 1 Dose Escalation Cohort: Mezagitamab 45 mg: Mezagitamab 45 mg, SC, once weekly for 8 weeks, then once every 2 weeks for 16 weeks, and then once every 4 weeks thereafter in a 28-day treatment cycle until progressive disease (PD), unacceptable toxicities or withdrawal due to other reasons.
Arm/Group | Phase 1 Dose Escalation Cohort: Mezagitamab 45 mg | Phase 1 Dose Escalation Cohort: Mezagitamab 135 mg | Phase 1 Dose Escalation Cohort: Mezagitamab 300 mg | Phase 1 Dose Escalation Cohort: Mezagitamab 600 mg | Phase 1 Dose Escalation Cohort: Mezagitamab 1200 mg | Phase 1 Combination Cohort: Mezagitamab 300 mg + PomDex
Number analyzed (Participants) | 4 | 3 | 12 | 22 | 3 | 6
hours (h)
  Cycle 1 Week 1 | 60.18 [22.88 to 168.00] | 70.60 [49.35 to 167.88] | 71.11 [44.00 to 168.50] | 72.55 [24.00 to 190.95] | 73.22 [70.23 to 169.30] | 70.58 [46.23 to 173.50]
  Cycle 2 Week 1: number analyzed (Participants) | 4 | 3 | 11 | 16 | 3 | 6
  Cycle 2 Week 1 | 58.77 [0.10 to 70.40] | 71.15 [22.78 to 168.57] | 70.00 [0 to 167.00] | 59.12 [0.25 to 172.53] | 71.92 [48.88 to 165.12] | 49.33 [5.67 to 70.85]

10. Secondary Outcome: AUClast: Area Under the Serum Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration for TAK-079
Time Frame: Cycle 1 and 2: Day 1 pre-dose and at multiple time points (up to 168 hours) post-dose (cycle length=28 days)
Population: PK analysis set included those participants from the safety analysis set who had sufficient dosing data and mezagitamab concentration-time data to permit the calculation of PK parameters. Overall number analyzed is the number of participants available for analyses. Number analyzed is the number of participants with data available for analysis at the given timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*nanogram/milliliter (h*ng/mL)
Arm/Group | Phase 1 Dose Escalation Cohort: Mezagitamab 45 mg | Phase 1 Dose Escalation Cohort: Mezagitamab 135 mg | Phase 1 Dose Escalation Cohort: Mezagitamab 300 mg | Phase 1 Dose Escalation Cohort: Mezagitamab 600 mg | Phase 1 Dose Escalation Cohort: Mezagitamab 1200 mg | Phase 1 Combination Cohort: Mezagitamab 300 mg + PomDex
Number analyzed (Participants) | 4 | 3 | 12 | 21 | 3 | 6
hours*nanogram/milliliter (h*ng/mL)
  Cycle 1 Week 1: number analyzed (Participants) | 2 | 3 | 12 | 21 | 3 | 6
  Cycle 1 Week 1 | 32800 (20.9) | 160000 (471.1) | 547000 (546.9) | 2710000 (83.8) | 5780000 (67.7) | 603000 (272.9)
  Cycle 2 Week 1: number analyzed (Participants) | 4 | 3 | 11 | 15 | 3 | 6
  Cycle 2 Week 1 | 10400 (285970.0) | 1920000 (159.8) | 4780000 (114.5) | 19300000 (79.6) | 27000000 (92.1) | 2690000 (33.9)

11. Secondary Outcome: Phase 1: Overall Response Rate (ORR)
Description: ORR is defined as the percentage of participants who achieved a partial response (PR) or better during the study. PR is defined as >=50% reduction of serum M-protein and reduction in 24-hour urinary M-protein by >=90% or to <200 mg/24 hours. If the serum and urine M-protein were not measurable, a ≥50% decrease in the difference between involved and uninvolved FLC levels was required in place of the M-protein criteria. If serum and urine M-protein were not measurable, and serum FLC was also not measurable, ≥50% reduction in bone marrow plasma cells was required in place of M-protein, provided the baseline percentage was ≥30%. In addition to the above criteria, if present at baseline, ≥50% reduction in the size of soft tissue plasmacytomas was also required. Two consecutive assessments were needed; no known evidence of progressive or new bone lesions if radiographic studies were performed. Percentages are rounded off to whole number at the nearest decimal.
Time Frame: Up to approximately 3.7 years
Population: Response-evaluable analysis set is a subset of the safety analysis set including participants with measurable disease at baseline and at least 1 posttreatment evaluation.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1 Dose Escalation Cohort: Mezagitamab 45 mg | Phase 1 Dose Escalation Cohort: Mezagitamab 135 mg | Phase 1 Dose Escalation Cohort: Mezagitamab 300 mg | Phase 1 Dose Escalation Cohort: Mezagitamab 600 mg | Phase 1 Dose Escalation Cohort: Mezagitamab 1200 mg | Phase 1 Combination Cohort: Mezagitamab 300 mg + PomDex
Number analyzed (Participants) | 4 | 3 | 12 | 19 | 3 | 6
percentage of participants | 25 [0.6 to 80.6] | 0 [0 to 0] | 42 [15.2 to 72.3] | 47 [24.4 to 71.1] | 33 [0.8 to 90.6] | 83 [35.9 to 99.6]

12. Secondary Outcome: Percentage of Participants With Minimal Response (MR)
Description: MR is defined as >=25% but <=49% reduction of serum M-protein and reduction in 24-hour urine M-protein by 50% to 89%. Percentages are rounded off to whole number at the nearest decimal.
Time Frame: Up to approximately 3.7 years
Population: as for outcome 11
Measure: Number; unit: percentage of participants
Arm/Group | Phase 1 Dose Escalation Cohort: Mezagitamab 45 mg | Phase 1 Dose Escalation Cohort: Mezagitamab 135 mg | Phase 1 Dose Escalation Cohort: Mezagitamab 300 mg | Phase 1 Dose Escalation Cohort: Mezagitamab 600 mg | Phase 1 Dose Escalation Cohort: Mezagitamab 1200 mg | Phase 1 Combination Cohort: Mezagitamab 300 mg + PomDex
Number analyzed (Participants) | 4 | 3 | 12 | 19 | 3 | 6
percentage of participants | 0 | 33 | 0 | 11 | 0 | 17

13. Secondary Outcome: Percentage of Participants With Positive Anti-drug Antibodies (ADA)
Description: Percentages are rounded off to whole number at the nearest decimal.
Time Frame: Up to approximately 3.7 years
Population: The immunogenicity analysis set included those participants from the safety population who had baseline and at least 1 postbaseline sample assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Phase 1 Dose Escalation Cohort: Mezagitamab 45 mg | Phase 1 Dose Escalation Cohort: Mezagitamab 135 mg | Phase 1 Dose Escalation Cohort: Mezagitamab 300 mg | Phase 1 Dose Escalation Cohort: Mezagitamab 600 mg | Phase 1 Dose Escalation Cohort: Mezagitamab 1200 mg | Phase 1 Combination Cohort: Mezagitamab 300 mg + PomDex
Number analyzed (Participants) | 2 | 1 | 12 | 18 | 3 | 6
percentage of participants | 0 | 0 | 8 | 0 | 0 | 17

14. Secondary Outcome: Phase 2a: Number of Participants With DLTs
Time Frame: From the first dose of study drug through 30 days after the last dose (up to approximately 3.7 years)
Population: as for outcome 7
Arm/Group | Phase 2a: Mezagitamab
Number analyzed (Participants) | 0

15. Secondary Outcome: Phase 2a: Number of Participants Reporting One or More TEAEs
Time Frame: From the first dose of study drug through 30 days after the last dose (up to approximately 3.7 years)
Population: as for outcome 7
Arm/Group | Phase 2a: Mezagitamab
Number analyzed (Participants) | 0

16. Secondary Outcome: Phase 2a: Number of Participants With TEAEs Leading to Dose Modifications
Time Frame: From the first dose of study drug through 30 days after the last dose (up to approximately 3.7 years)
Population: as for outcome 7
Arm/Group | Phase 2a: Mezagitamab
Number analyzed (Participants) | 0

17. Secondary Outcome: Phase 2a: Number of Participants With TEAEs Leading to Treatment Discontinuation
Time Frame: From the first dose of study drug through 30 days after the last dose (up to approximately 3.7 years)
Population: as for outcome 7
Arm/Group | Phase 2a: Mezagitamab
Number analyzed (Participants) | 0

18. Secondary Outcome: Phase 2a: Duration of Response (DOR)
Description: DOR is the time from date of first documentation of response to date of first documented PD. PD is increase of >=25% from lowest response value in any of following:Serum M-protein(increase must be >=0.5 gram per deciliter[g/dL];serum M component increases >=1 g/dL are sufficient to define relapse if starting M component is >=5 g/dL),and/or urine M-protein(increase must be >=200 mg/24 hour), and/or only in participants without measurable serum and urine M-protein levels, difference between involved/uninvolved FLC levels (increase must be >10 mg/dL), and only in participants without measurable serum and urine M-protein levels and without measurable disease by FLC levels, bone marrow plasma cell percentage (percentage must be >=10%) or definite development of new bone lesions or soft tissue plasmacytomas or increase in size of bone lesions or soft tissue plasmacytomas, and development of hypercalcemia that can be attributed solely to plasma cell proliferative disorder.
Time Frame: Up to approximately 3.7 years
Population: as for outcome 7
Arm/Group | Phase 2a: Mezagitamab
Number analyzed (Participants) | 0

19. Secondary Outcome: Phase 2a: Progression Free Survival (PFS)
Description: PFS is time from the date of the first dose until the earliest date of disease progression (PD). PD is increase of >=25% from lowest response value in any of following: Serum M-protein (increase must be >=0.5 g/dL; serum M component increases >=1 g/dL are sufficient to define relapse if starting M component is >=5 g/dL),and/or urine M-protein (increase must be >=200 mg/24 hour), and/or only in participants without measurable serum and urine M-protein levels, difference between involved/uninvolved FLC levels (increase must be >10 mg/dL), and only in participants without measurable serum and urine M-protein levels and without measurable disease by FLC levels, bone marrow plasma cell percentage (percentage must be >=10%) or definite development of new bone lesions or soft tissue plasmacytomas or increase in size of bone lesions or soft tissue plasmacytomas, and development of hypercalcemia that can be attributed solely to plasma cell proliferative disorder.
Time Frame: Up to approximately 3.7 years
Population: as for outcome 7
Arm/Group | Phase 2a: Mezagitamab
Number analyzed (Participants) | 0

20. Secondary Outcome: Phase 2a: Overall Survival (OS)
Description: OS is defined as the time from the date of first dose to the date of death due to any cause.
Time Frame: Up to approximately 3.7 years
Population: as for outcome 7
Arm/Group | Phase 2a: Mezagitamab
Number analyzed (Participants) | 0

21. Secondary Outcome: Phase 2a: Time to Response (TTR)
Description: TTR is defined as the time from the date of the first dose to the date of the first documentation of response (PR [partial response] or better). PR is defined as >=50% reduction of serum M-protein and reduction in 24-hour urinary M-protein by >=90% or to <200 mg/24 hours.
Time Frame: Up to approximately 3.7 years
Population: as for outcome 7
Arm/Group | Phase 2a: Mezagitamab
Number analyzed (Participants) | 0

22. Secondary Outcome: Phase 1: RP2D of TAK-079
Description: RP2D was determined by dose escalating monotherapy groups.
Time Frame: From the first dose of study drug through 30 days after the last dose (up to approximately 3.7 years)
Population: as for outcome 2
Measure: Number; unit: mg
Groups:
- Phase 1 Dose Escalation Cohort: Mezagitamab: Mezagitamab SC, at escalating doses ranging from 45 mg to 1200 mg once weekly for 8 weeks, then once every 2 weeks for 16 weeks, and then once every 4 weeks thereafter in a 28-day treatment cycle until PD, unacceptable toxicities or withdrawal due to other reasons.
Arm/Group | Phase 1 Dose Escalation Cohort: Mezagitamab
Number analyzed (Participants) | 37
mg | 600

ADVERSE EVENTS:
Time Frame: From the first dose of study drug through 30 days after the last dose (up to approximately 3.7 years)
Description: At each visit the investigator documented any occurrence of adverse events and clinically significant abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment. Safety analysis set included all enrolled participants who received at least 1 dose of study drug.
Arm/Group | Phase 1 Dose Escalation Cohort: Mezagitamab 45 mg | Phase 1 Dose Escalation Cohort: Mezagitamab 135 mg | Phase 1 Dose Escalation Cohort: Mezagitamab 300 mg | Phase 1 Dose Escalation Cohort: Mezagitamab 600 mg | Phase 1 Dose Escalation Cohort: Mezagitamab 1200 mg | Phase 1 Combination Cohort: Mezagitamab 300 mg + PomDex
All-Cause Mortality (participants affected / at risk) | 1/4 | 0/3 | 7/12 | 6/22 | 1/3 | 1/6
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/3 | 1/12 | 8/22 | 1/3 | 2/6
Other Adverse Events (participants affected / at risk) | 4/4 | 3/3 | 12/12 | 21/22 | 3/3 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1 Dose Escalation Cohort: Mezagitamab 45 mg (N=4) | Phase 1 Dose Escalation Cohort: Mezagitamab 135 mg (N=3) | Phase 1 Dose Escalation Cohort: Mezagitamab 300 mg (N=12) | Phase 1 Dose Escalation Cohort: Mezagitamab 600 mg (N=22) | Phase 1 Dose Escalation Cohort: Mezagitamab 1200 mg (N=3) | Phase 1 Combination Cohort: Mezagitamab 300 mg + PomDex (N=6)
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Soft tissue infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1 Dose Escalation Cohort: Mezagitamab 45 mg (N=4) | Phase 1 Dose Escalation Cohort: Mezagitamab 135 mg (N=3) | Phase 1 Dose Escalation Cohort: Mezagitamab 300 mg (N=12) | Phase 1 Dose Escalation Cohort: Mezagitamab 600 mg (N=22) | Phase 1 Dose Escalation Cohort: Mezagitamab 1200 mg (N=3) | Phase 1 Combination Cohort: Mezagitamab 300 mg + PomDex (N=6)
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 3 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 3 | 4 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 1 | 2 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 1 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4 | 5 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 2 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 2 | 0 | 0
Blood pressure increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0
Bruxism (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1 | 0 | 0
Chills (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 0 | 2
Coronavirus test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 2 | 0 | 2
Cranial nerve paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 2 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 1 | 3 | 1 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 1 | 0 | 0 | 1
Dyskinesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 2 | 1 | 1
Early satiety (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 4 | 5 | 2 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 1
Folliculitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Fungal skin infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 1
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 4 | 2 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 1 | 1 | 0 | 4 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Injection site haemorrhage (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1 | 3 | 5 | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 2 | 0 | 1 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 1 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 3 | 3 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 2 | 1 | 3
Neutrophil count decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 3
Nocturia (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 1 | 0 | 0
Oedema (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 4 | 0 | 0
Oesophageal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 1 | 1 | 0 | 0
Peripheral swelling (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 1 | 1 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 3 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 2 | 0 | 0
Rash follicular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Soft tissue infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 0 | 0
Tongue ulceration (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 2 | 7 | 1 | 2
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 2
Varicose vein (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Venous thrombosis limb (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 1 | 1 | 0 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.

DOCUMENTS (2):
  • Study Protocol (2019-04-02): https://cdn.clinicaltrials.gov/large-docs/80/NCT03439280/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-11): https://cdn.clinicaltrials.gov/large-docs/80/NCT03439280/SAP_001.pdf